CLINICAL TRIAL: NCT05549817
Title: Synchronous and Asynchronous Telerehabilitation Methods in Patients With Shoulder Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/67
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Tendinopathy; Shoulder Pain
MeSH Terms: conditions — Tendinopathy; Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation Group (Experimental): The exercise program was applied to groups that include three participants of the synchronous group 3 days per week by video conference method on an online platform (Zoom) with the supervision of a physiotherapist. The time of the group session was organized according to the availability of participants in that group and the physiotherapist using shared calendar availability (Doodle). The physiotherapist sent a reminder to participants one hour prior to each session including the video conference meeting link. Each exercise session lasted approximately 40 minutes. For 8 weeks, a total of 24 exercise sessions were performed. The physiotherapist demonstrated the exercises as needed, supervised the group by giving real-time feedback, and progressed the exercise program according to the needs of each group.
  Interventions: Other: Synchronous Exercise Program
- Asynchronous Telerehabilitation Group (Active Comparator): The exercise program was prescribed and followed up 3 days per week via the mobile application (FizyoTr). A notification was sent to participants' phones via mobile application prior to each session and attendance to the exercise program was recorded. For 8 weeks, a total of 24 exercise sessions were performed. The physiotherapist progressed the exercise program according to the assessment at 4 weeks and the needs of each participant.
  Interventions: Other: Asynchronous Exercise Program

INTERVENTIONS:
Other: Synchronous Exercise Program — The exercise program consisted of exercises by recommended guidelines for shoulder tendinopathy patients which includes various strengthening, stretching, and proprioceptive exercises with progression.
  Arms: Synchronous Telerehabilitation Group
Other: Asynchronous Exercise Program — The exercise program consisted of exercises by recommended guidelines for shoulder tendinopathy patients which includes various strengthening, stretching, and proprioceptive exercises with progression.
  Arms: Asynchronous Telerehabilitation Group

SUMMARY:
This study is a randomized controlled trial conducted to compare the effects of synchronous and asynchronous telerehabilitation programs on pain, disability, and quality of life parameters in patients with shoulder tendinopathy in the Marmara University Physiotherapy and Rehabilitation Department.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18-65,
* Who had access to the internet and smartphone,
* Had the ability to conduct video calls included in the study.

Exclusion Criteria:

* Participants were excluded if they had COVID-19,
* Had surgery in the last 6 months,
* Had neurological and psychological disorders,
* Received physiotherapy treatment.
* Had surgery in the last 6 months,
* Had a condition that prevented them from exercising.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | The pain was measured at baseline.
  Pain intensity was measured with a 0-10 cm scale. Participants were asked to rate their pain as "0: no pain and 10: excruciating pain" on the 0-10 cm scale (10). The pain reported by the patients was recorded in centimeters.
Numerical Pain Rating Scale (NPRS) | The pain was measured at mid-treatment in the 4th week.
  Pain intensity was measured with a 0-10 cm scale. Participants were asked to rate their pain as "0: no pain and 10: excruciating pain" on the 0-10 cm scale (10). The pain reported by the patients was recorded in centimeters.
Numerical Pain Rating Scale (NPRS) | The pain was measured at the end of treatment in the 8th week.
  Pain intensity was measured with a 0-10 cm scale. Participants were asked to rate their pain as "0: no pain and 10: excruciating pain" on the 0-10 cm scale (10). The pain reported by the patients was recorded in centimeters.
Numerical Pain Rating Scale (NPRS) | The pain was measured at long-term follow-up assessment in the 16th week.
  Pain intensity was measured with a 0-10 cm scale. Participants were asked to rate their pain as "0: no pain and 10: excruciating pain" on the 0-10 cm scale (10). The pain reported by the patients was recorded in centimeters.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | The disability was measured at baseline.
  The DASH survey was published in 1994 by the American Academy of Orthopedic Developed by Surgeons (AAOS), in upper extremity injuries. It is a questionnaire that evaluates function and disability. The survey consists of 30 questions. The first 21 questions about the difficulty of the patient during activities of daily living, 5 questions about symptoms (pain, activity-related pain, tingling, stiffness, weakness), social function, work, sleep, and patient self-esteem in each of the remaining 4 questions. A total score of 0-100 is obtained. High scores indicate severe disability (0 points: no disability, 100 points: maximum disability). Turkish validity and reliability study of the survey was conducted.
Disabilities of the Arm, Shoulder and Hand (DASH) | The disability was measured at mid-treatment in the 4th week.
  The DASH survey was published in 1994 by the American Academy of Orthopedic Developed by Surgeons (AAOS), in upper extremity injuries. It is a questionnaire that evaluates function and disability. The survey consists of 30 questions. The first 21 questions about the difficulty of the patient during activities of daily living, 5 questions about symptoms (pain, activity-related pain, tingling, stiffness, weakness), social function, work, sleep, and patient self-esteem in each of the remaining 4 questions. A total score of 0-100 is obtained. High scores indicate severe disability (0 points: no disability, 100 points: maximum disability). Turkish validity and reliability study of the survey was conducted.
Disabilities of the Arm, Shoulder and Hand (DASH) | The disability was measured at the end of treatment in the 8th week.
  The DASH survey was published in 1994 by the American Academy of Orthopedic Developed by Surgeons (AAOS), in upper extremity injuries. It is a questionnaire that evaluates function and disability. The survey consists of 30 questions. The first 21 questions about the difficulty of the patient during activities of daily living, 5 questions about symptoms (pain, activity-related pain, tingling, stiffness, weakness), social function, work, sleep, and patient self-esteem in each of the remaining 4 questions. A total score of 0-100 is obtained. High scores indicate severe disability (0 points: no disability, 100 points: maximum disability). Turkish validity and reliability study of the survey was conducted.
Disabilities of the Arm, Shoulder and Hand (DASH) | The disability was measured at long-term follow-up assessment in the 16th week.
  The DASH survey was published in 1994 by the American Academy of Orthopedic Developed by Surgeons (AAOS), in upper extremity injuries. It is a questionnaire that evaluates function and disability. The survey consists of 30 questions. The first 21 questions about the difficulty of the patient during activities of daily living, 5 questions about symptoms (pain, activity-related pain, tingling, stiffness, weakness), social function, work, sleep, and patient self-esteem in each of the remaining 4 questions. A total score of 0-100 is obtained. High scores indicate severe disability (0 points: no disability, 100 points: maximum disability). Turkish validity and reliability study of the survey was conducted.
Short Form-36 (SF-36) | The quality of life was measured at baseline.
  The quality of life was assessed using SF-36, which consists of 36 items. The Sf-36 has a total of 8 subscales including physical functioning, limitation due to physical problems (physical role), limitation due to emotional problems (emotional role), vitality, bodily pain, mental health, general health, and social functioning. The Turkish version of the SF-36 has been shown to have validity and reliability.
Short Form-36 (SF-36) | The quality of life was measured at mid-treatment in the 4th week.
  The quality of life was assessed using SF-36, which consists of 36 items. The Sf-36 has a total of 8 subscales including physical functioning, limitation due to physical problems (physical role), limitation due to emotional problems (emotional role), vitality, bodily pain, mental health, general health, and social functioning. The Turkish version of the SF-36 has been shown to have validity and reliability.
Short Form-36 (SF-36) | The quality of life was measured at the end of treatment in the 8th week.
  The quality of life was assessed using SF-36, which consists of 36 items. The Sf-36 has a total of 8 subscales including physical functioning, limitation due to physical problems (physical role), limitation due to emotional problems (emotional role), vitality, bodily pain, mental health, general health, and social functioning. The Turkish version of the SF-36 has been shown to have validity and reliability.
Short Form-36 (SF-36) | The quality of life was measured at long-term follow-up assessment in the 16th week.
  The quality of life was assessed using SF-36, which consists of 36 items. The Sf-36 has a total of 8 subscales including physical functioning, limitation due to physical problems (physical role), limitation due to emotional problems (emotional role), vitality, bodily pain, mental health, general health, and social functioning. The Turkish version of the SF-36 has been shown to have validity and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No